CLINICAL TRIAL: NCT00825617
Title: Quantitative Liver Functions in Turner Syndrome With and Without Hormone Replacement Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: MD, PhD, DMSc Claus H. Gravholt, Medical department M, Aarhus University Hospital, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19963561
Record Dates: First submitted 2009-01-20; First posted 2009-01-21 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Turner Syndrome
Keywords: TS; HRT; Liver function tests
MeSH Terms: conditions — Turner Syndrome | interventions — Hormone Replacement Therapy; Trisequens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HRT (Experimental): Women with TS were treated with oral hormone substitution consisting of 2 mg 17β-estradiol/day for days 1-12, 2 mg 17β-estradiol/day and 1 mg norethisterone acetate/day for days 13-22 and 1 mg 17β-estradiol/day for days 23-28 (Trisekvens, Novo Nordisk A/S, Bagsværd, Denmark)
  Interventions: Drug: Hormone replacement therapy

INTERVENTIONS:
Drug: Hormone replacement therapy — Women with TS were treated with oral hormone substitution consisting of 2 mg 17β-estradiol/day for days 1-12, 2 mg 17β-estradiol/day and 1 mg norethisterone acetate/day for days 13-22 and 1 mg 17β-estradiol/day for days 23-28 (Trisekvens, Novo Nordisk A/S, Bagsværd, Denmark)
  Other Names: Trisekvens, Novo Nordisk A/S, Bagsværd, Denmark

SUMMARY:
Several studies have demonstrated that Turner Syndrome patients have elevated liver enzymes readily suppressible by a short course of HRT. We wanted to estimated quantitative liver functions in a young group of Turner syndrome patients compared to a healthy control group.

DETAILED DESCRIPTION:
Turner syndrome is due to the absence of a part of or the entire X chromosome in females. Stature is short, and morbidity is increased due to risk of osteoporosis and fractures, type 2 diabetes, ischemic heart disease, hypertension, and stroke, but also the risk of cirrhosis is increased. Clinical studies have shown a frequent occurrence of elevated liver enzymes, primarily alanine aminotransferase, g-glutamyl-transferase, and alkaline phosphatase, while bilirubin is normal.

We and others have shown a normalizing effect of hormone replacement therapy (HRT), containing 17bestradiol and a gestagen, on liver enzymes, which may point towards a protective effect on hepatocyte integrity. Marked architectural changes, including nodular regenerative hyperplasia, multiple focal nodular hyperplasia and cirrhosis are observed in some patients and are associated with a risk of liver-related complications. These changes are frequently associated with vascular disorders such as obliterative portal venopathy, probably related to congenitally abnormal vessels. Steatosis, steatofibrosis, and steatohepatitis are seen and may be caused by metabolic disorders. In addition, bile duct alterations resembling small duct sclerosing cholangitis are observed in several patients. Presently, it is not known whether these perturbations in liver morphology and in liver-derived enzymes are related to functional defects in females with TS and whether this may change by HRT. To further explore quantitative liver function in TS, we examined adult women with TS on and off HRT and compared them with a control group of age matched normal women. We used the galactose elimination capacity to assess hepatocyte cytosol activity, the plasma clearance of indocyanine green to assess hepatic blood flow and excretory liver cell function independently of hepatic blood flow, the antipyrine plasma clearance to estimate hepatic microsomal system activity, and the functional hepatic nitrogen clearance to assess mitochondrial- cytosolic metabolic capacity for conversion of amino-nitrogen.We assumed that one or more these metabolic liver functions would be diminished in untreated TS and normalized by HRT. Our principal objective was to understand mechanistically how HRT improves liver function in TS.

ELIGIBILITY:
Inclusion Criteria:

* Turner syndrome by karyotype

Exclusion Criteria:

* Thyroid abnormality
* Glucocorticoid treatment

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 1996-10; Primary Completion 1999-10 (Actual); Study Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
quantitative liver function tests | 1996-1999

CONTACTS AND LOCATIONS:
Overall Officials: J S Christíansen, Professor, Principal Investigator — Medical departmnet M, Aarhus University Hospital, NBG, Denamrk,
Locations (1):
- Medical department M and Investigational Laboratories, Aarhus C, Jutland, Denmark